CLINICAL TRIAL: NCT06879106
Title: Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Brief Title: Effect of Cognitive Therapy on Immunosuppressive Treatment Compliance and Motivation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: okutan8
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Liver Transplant; Complications; Immunosuppression; Compliance, Treatment
Keywords: Mindfulness-Based Cognitive Therapy (MBCT); liver transplantation; immunosuppressive therapy; compliance; motivation level
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pretestpost- test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Data collection tools will be applied to the patients in the experimental group before the MBCT intervention. The 60 patients in the experimental group will be divided into six subgroups of 10 patients each. During the MBCT intervention, eight consecutive sessions will be held with the themes of "Mindfulness and Autopilot", "Living in Our Mind", "Focusing on the Distracted Mind", "Recognizing Hate", "Allowing", "Thoughts Are Not Real", "How Can I Best Take Care of Myself?" and "Maintaining and Expanding New Learning". One MBCT session will be held per week and therefore the MBCT program will continue for eight weeks. After the eight-week MBCT program ends, no intervention will be applied to the patients in the experimental group for the next month based on similar studies in the literature and at the end of this one month, in the posttest phase, these patients will be applied the scales once more.
  Interventions: Other: Intervention group
- control group (No Intervention): Control group Data collection tools will be applied to patients in the control group as part of the pre-test. Patients with questions will be allowed to direct their questions to the researchers. After these questions are answered, no intervention will be made to the control group and patients in the control group will not be contacted at any time for the next three months. After three months, patients in the control group will be invited to the outpatient clinic and the scales will be applied to these patients once more during these outpatient clinic visits to collect post-test data.

INTERVENTIONS:
Other: Intervention group — The Mindfulness-Based Cognitive Therapy (MBCT) intervention is an educational program consisting of the themes "Mindfulness and Autopilot," "Living in Our Mind," "Focusing the Distracted Mind," "Recognizing Hate," "Allowing," "Thoughts Are Not Real," "How Can I Best Take Care of Myself," and "Sustaining and Expanding New Learning."
  Arms: Intervention group

SUMMARY:
The study aims to analyze the effects of Mindfulness-Based Cognitive Therapy (MBCT) on the motivation levels and compliance with immunosuppressive therapy of post-liver transplant recipients.

H1-0: MBCT has no effect on the compliance of recipients to immunosuppressive therapy after liver transplantation.

H1-1: MBCT has an effect on the compliance of recipients to immunosuppressive therapy after liver transplantation.

H2-0: MBCT has no effect on increasing the motivation of recipients after liver transplantation.

H2-1: MBCT has an effect on increasing the motivation of recipients after liver transplantation.

DETAILED DESCRIPTION:
Experimental group Data collection tools will be applied to the patients in the experimental group before the MBCT intervention. The 60 patients in the experimental group will be divided into six subgroups, each consisting of 10 patients. MBCT will be applied by Expert Clinical Psychologist Aybüke İğdir, who has received special training in the field. There will be a group facilitator among the MBCT trainers. The group facilitator is a psychologist with postgraduate education and experience in MBCT. The MBCT intervention will be applied to each subgroup of the experimental group on different days. During the MBCT intervention, eight consecutive sessions will be held with the themes of "Mindfulness and Autopilot", "Living in Our Mind", "Focusing on the Distracted Mind", "Recognizing Hate", "Allowing", "Thoughts Are Not Real", "How Can I Best Take Care of Myself?" and "Maintaining and Expanding New Learning". The theme of Maintaining and Expanding New Learning includes special techniques that patients can apply for medication compliance. There will be one MBCT session per week and therefore the MBCT program will continue for eight weeks. After the eight-week MBCT program ends, no intervention will be applied to the patients in the experimental group for the next month based on similar studies in the literature and at the end of this one month, in the posttest phase, these patients will be applied the scales once again.

Control group Data collection tools will be applied to patients in the control group as part of the pre-test. Patients with questions will be allowed to direct their questions to the researchers. After these questions are answered, no intervention will be made to the control group and patients in the control group will not be contacted at any time for the next three months. After three months, patients in the control group will be invited to the outpatient clinic and the scales will be applied to these patients once more during these outpatient clinic visits to collect post-test data.

ELIGIBILITY:
Inclusion Criteria:

* Applying to the outpatient clinic for routine follow-up after liver transplantation,
* Receiving immunosuppressive treatment for at least one month after liver transplantation,
* Being 18 years old or older,
* Not having a communication barrier,
* Agreeing to participate in the study.

Exclusion Criteria:

* Having any hearing or mental problems
* Wanting to leave the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to Immunosuppressive Therapy | It will take approximately 5 minutes
  Immunosuppressant Therapy Adherence Scale (ITAS) This scale was first developed in 1986 by Morisky and colleagues to assess the adherence of hypertensive patients to anti-hypertensive drugs. It consists of four items, each of which assesses how many times and why the recipient forgot to take immunosuppressive drugs to prevent transplant rejection in the last three months. In scoring, participants who fully adhered to immunosuppressive drug treatment in the last three months were given 3 points, those with a non-adherence rate of 1-20% were given 2 points, those with a non-adherence rate of 21-50% were given 1 point, and those with a non-adherence rate of more than 50% were given 0 points. A participant can score between 0 and 12 on the ITAS. A high ITAS score indicates a high level of adherence to treatment.
Mindful Attention | It will take approximately 15 minutes
  Mindful Attention Scale (MAAS) MAAS was created by Brown and Ryan and is used to measure the awareness levels of individuals. It is a six-point Likert-type scale consisting of 15 items and is evaluated based on a single total score. A high MAAS score indicates that the participant has a high level of awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, PhD., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)